CLINICAL TRIAL: NCT00613938
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Tapentadol Immediate-Release Formulation in the Treatment of Acute Pain From Bunionectomy
Brief Title: A Study to Evaluate the Effectiveness and Safety of Tapentadol (CG5503) in the Treatment of Acute Pain From Bunionectomy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014116; KF5503/38
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-04-23 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Arthralgia; Bunion; Hallux Valgus; Pain
Keywords: Acute pain; bunionectomy; tapentadol
MeSH Terms: conditions — Arthralgia; Bunion; Hallux Valgus; Pain; Acute Pain | interventions — Tapentadol; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 004 (Placebo Comparator): placebo 1 capsule q4-6 hrs for 3 days
  Interventions: Drug: placebo
- 003 (Active Comparator): oxycodone 10mg capsule q4-6 hrs for 3 days
  Interventions: Drug: oxycodone
- 001 (Experimental): Tapentadol (CG5503) 50mg capsule q4-6 hrs for 3 days
  Interventions: Drug: Tapentadol (CG5503)
- 002 (Experimental): Tapentadol (CG5503) 75mg capsule q4-6 hrs for 3 days
  Interventions: Drug: Tapentadol (CG5503)

INTERVENTIONS:
Drug: Tapentadol (CG5503) — 50mg capsule q4-6 hrs for 3 days
  Arms: 001
Drug: Tapentadol (CG5503) — 75mg capsule q4-6 hrs for 3 days
  Arms: 002
Drug: oxycodone — 10mg capsule q4-6 hrs for 3 days
  Arms: 003
Drug: placebo — 1 capsule q4-6 hrs for 3 days
  Arms: 004

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of 2 different dose levels of tapentadol (CG5503) compared with oxycodone and with placebo in subjects who have had a bunionectomy.

DETAILED DESCRIPTION:
Patients undergoing bunionectomy often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when patients receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, and less frequently, respiratory depression. Tapentadol (CG5503), a newly synthesized drug with an immediate release (IR) formulation, also acts as a centrally acting analgesic but has a dual mode of action. The aim of this study is to investigate the effectiveness (level of pain control) and safety (side effects) of 2 dose levels of tapentadol (CG5503) IR compared to no drug (placebo) or one dose level of oxycodone (an opioid commonly used to treat post-surgical pain). This study is a randomized, double-blind (neither investigator nor patient will know which treatment is received), active- and placebo-controlled, parallel-group, multicenter study to evaluate treatment of the acute pain from bunionectomy. The study will include a blinded 72 hour inpatient (the patient will stay in the facility where the procedure is done) phase immediately following bunionectomy, during which patients will be treated with either 50- or 75-mg tapentadol (CG5503) IR, a placebo, or 10-mg oxycodone IR, and pain relief will be periodically assessed. Assessments of pain intensity (PI) and pain relief (PAR) are obtained using the numerical rating scale, and the patient global impression of change scale (PGIC) will measure overall patient status. Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of tapentadol (CG5503) and oxycodone. The study hypotheses are that at least one tapentadol (CG5503) IR dose will be different from placebo in controlling patients pain at 48 hours, followed by establishing that at least one tapentadol (CG5503) IR dose will be non-inferior compared with oxycodone IR (oxycodone IR is not clinically significantly better than a tapentadol (CG5503) IR dose). A comparison of the incidence rate of the adverse events of nausea and/or vomiting, and the incidence rate of the adverse event of constipation, between tapentadol (CG5503) IR and oxycodone IR will also be performed. Tapentadol (CG5503) IR 50 or 75 mg, or oxycodone 10 mg, or placebo, 1 capsule taken by mouth every 4 to 6 hours during the 72-hour postsurgery phase of the study (acetaminophen is also allowed during the first 12 hours on Day 1, if needed for pain). All doses of study treatment will be taken with approximately 120 mL of water with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Patients must undergo primary unilateral first metatarsal bunionectomy
* Pain intensity must be moderate to severe following removal of a continuous popliteal sciatic block
* Female patients must be postmenopausal, surgically sterile, or practicing an effective method of birth control if they are sexually active.

Exclusion Criteria:

* Patients will be excluded from the study if they have a history of seizure disorder or epilepsy
* History of malignancy within the past 2 years before starting the study
* History of alcohol or drug abuse
* Evidence of active infections that may spread to other areas of the body
* Clinical laboratory values reflecting severe renal insufficiency
* Moderately or severely impaired hepatic function
* Currently treated with anticonvulsants, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), neuroleptics, or serotonin norepinephrine reuptake inhibitor (SNRI).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (7):
- United States (7):
  - Glendale, California
  - Pasadena, Maryland
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - San Marcos, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Daniels S, Casson E, Stegmann JU, Oh C, Okamoto A, Rauschkolb C, Upmalis D. A randomized, double-blind, placebo-controlled phase 3 study of the relative efficacy and tolerability of tapentadol IR and oxycodone IR for acute pain. Curr Med Res Opin. 2009 Jun;25(6):1551-61. doi: 10.1185/03007990902952825. PMID 19445652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this inpatient, multicenter study occurred between January 28, 2008 and October 3, 2008.
Pre-assignment Details: The study consisted of a screening period (duration up to 28 days), and a double blind active treatment period (4 days).
Groups:
- Placebo: Placebo capsule taken by mouth every 4 to 6 hours for 3 days.
- Tapentadol 50mg Fixed Dose: Tapentadol 50mg capsule taken by mouth every 4 to 6 hours for 3 days.
- Tapentadol 75mg Fixed Dose: Tapentadol 75mg capsule taken by mouth every 4 to 6 hours for 3 days.
- Oxycodone 10mg Fixed Dose: Oxycodone 10mg capsule taken by mouth every 4 to 6 hours for 3 days.
Period: Overall Study
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Started | 69 | 275 | 278 | 279 (one patient did not have a valid baseline score therefore excluded from above)
Completed | 49 | 247 | 255 | 253
Not Completed | 20 | 28 | 23 | 26
Not completed — Withdrawal by Subject | 2 | 4 | 9 | 9
Not completed — Adverse Event | 1 | 4 | 8 | 5
Not completed — Lack of Efficacy | 16 | 18 | 5 | 9
Not completed — Other | 1 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose | Total
Number analyzed (Participants) | 69 | 275 | 278 | 279 | 901
Age, Categorical [Number; unit: participants] — One patient in the oxycodone 10mg group did not have a valid baseline score and was therefore excluded from the safety analysis set.
  participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 68 | 265 | 268 | 265 | 866
    >=65 years | 1 | 10 | 10 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.65) | 42.4 (13.23) | 43.5 (12.57) | 43.4 (13.25) | 43.1 (13.05)
Gender [Number; unit: participants] — One patient in the oxycodone 10mg group did not have a valid baseline score and was therefore excluded from the safety analysis set.
  participants
    Female | 64 | 232 | 248 | 233 | 777
    Male | 5 | 43 | 30 | 45 | 123
Region of Enrollment [Number; unit: participants] — One patient in the oxycodone 10mg group did not have a valid baseline score and was therefore excluded from the safety analysis set.
  participants
    United States | 69 | 275 | 278 | 278 | 900

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference Over 48 Hours (SPID48)
Description: The SPID score incorporates the cumulative analgesic effects of tapentadol IR on pain intensity over an extended period (48 hours) allowing for an evaluation of multiple doses of drug, even when dosing frequency may vary. Scoring is derived from the Numerical Rating Scale (NRS) from 0 = No pain to 11 = Pain as bad as you can imagine. A positive difference between the mean SPID48 for an active study drug and placebo would indicate a numerically larger analgesic effect for subjects dosed with active study drug than in the placebo group. A higher value in SPID indicates greater pain relief.
Time Frame: 48 hours
Population: The primary analysis set was the Intent to Treat (ITT) analysis set that included all subjects who were randomized, received at least one dose of study drug and had a non-missing baseline pain intensity score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 69 | 275 | 278 | 278
Scores on a scale | 54.1 (105.74) | 122.2 (98.66) | 143.7 (96.52) | 140.3 (99.52)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol 50mg Fixed Dose vs Tapentadol 75mg Fixed Dose vs Oxycodone 10mg Fixed Dose; Null hypothesis: There are no differences in pain intensity measured by SPID-48 hours between any of tapentadol dose groups and placebo. ANCOVA model with factors of treatment, center and baseline pain intensity score was used for the primary analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparisons of tapentadol dose groups and placebo was performed with Hochberg procedure for adjustment for the multiple tests; Mean Difference (Final Values) = 62.4, 95% CI [39.01 to 85.73], Standard Error of Mean 11.9 — The results shown are the treatment group differences between Tapentadol IR 50mg group and placebo

2. Secondary Outcome: Time to First Rescue Pain Medication Use.
Description: The effect of tapentadol (CG5503) IR on the time to the first use of rescue pain medication.
Time Frame: 3 days
Population: as for outcome 1
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: The SPID at 12 Hours Relative to First Dose.
Description: The SPID score incorporates the cumulative analgesic effects of tapentadol IR on pain intensity over an extended period (12 to 72 hours) allowing for an evaluation of multiple doses of drug, even when dosing frequency may vary. Scoring is derived from the Numerical Rating Scale (NRS) from 0 = No pain to 11 = Pain as bad as you can imagine. A positive difference between the mean SPID12 for an active study drug and placebo would indicate a numerically larger analgesic effect for subjects dosed with active study drug than in the placebo group. A higher value in SPID indicates greater pain relief.
Time Frame: 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 69 | 275 | 278 | 278
Scores on a scale | 7.5 (20.7) | 21.1 (21.89) | 26.0 (23.11) | 24.9 (22.8)

4. Secondary Outcome: SPID at 24 Hours Relative to First Dose
Description: The SPID score incorporates the cumulative analgesic effects of tapentadol IR on pain intensity over an extended period (12 to 72 hours) allowing for an evaluation of multiple doses of drug, even when dosing frequency may vary. Scoring is derived from the Numerical Rating Scale (NRS) from 0 = No pain to 11 = Pain as bad as you can imagine. A positive difference between the mean SPID24 for an active study drug and placebo would indicate a numerically larger analgesic effect for subjects dosed with active study drug than in the placebo group. A higher value in SPID indicates greater pain relief.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 69 | 275 | 278 | 278
Scores on a scale | 12.1 (43.64) | 45.4 (45.73) | 58.1 (45.89) | 53.8 (46.69)

5. Secondary Outcome: Percentage of Patients Who Reported Very Much Improved or Much Improved From Baseline in Patient Global Impression of Change to Day 3
Description: Ordinal measure indicating change from the start of treatment (On a scale of 7 = Very much Worse to 1 = very much improved) to endpoint at Day 3
Time Frame: Baseline and 3 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 69 | 275 | 278 | 278
percentage of participants | 65.2 | 83.2 | 87.8 | 86.0

6. Secondary Outcome: Total Pain Relief (TOTPAR)at 48 Hours
Description: Total Pain Relief (TOTPAR48) was defined as the weighted sum over all pain relief scores(PAR) from 0.5 hour to Hour 48, with the actual time elapsed from the previous PAR observation as the weight. A higher value in TOTPAR indicates greater pain relief.
Time Frame: 48 hours
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Number analyzed (Participants) | 69 | 275 | 278 | 278
scores on a scale | 68.2 (39.48) | 96.6 (37.39) | 107.5 (35.74) | 105.2 (37.4)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded from the time that the informed consent (ICF) was obtained until the last study procedure had been completed. For subjects who discontinued early, AEs were collected for 48 hours after the last intake of study drug.
Arm/Group | Placebo | Tapentadol 50mg Fixed Dose | Tapentadol 75mg Fixed Dose | Oxycodone 10mg Fixed Dose
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/275 | 0/278 | 1/279
Other Adverse Events (participants affected / at risk) | 25/69 | 161/275 | 192/278 | 218/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=69) | Tapentadol 50mg Fixed Dose (N=275) | Tapentadol 75mg Fixed Dose (N=278) | Oxycodone 10mg Fixed Dose (N=279)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=69) | Tapentadol 50mg Fixed Dose (N=275) | Tapentadol 75mg Fixed Dose (N=278) | Oxycodone 10mg Fixed Dose (N=279)
Alanine aminotransferase increased (Investigations) | 1 | 8 | 7 | 14
Constipation (Gastrointestinal disorders) | 1 | 22 | 15 | 31
Dizziness (Nervous system disorders) | 7 | 41 | 69 | 65
Headache (Nervous system disorders) | 11 | 56 | 52 | 73
Nausea (Gastrointestinal disorders) | 12 | 93 | 127 | 160
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 14 | 23 | 28
Somnolence (Nervous system disorders) | 2 | 20 | 37 | 33
Vomiting (Gastrointestinal disorders) | 0 | 34 | 77 | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days